CLINICAL TRIAL: NCT05328791
Title: Effectiveness of a Mindfulness Based Diet Program Given to Obese Individuals on Body Weight and Eating Behaviours
Brief Title: Effectiveness of a Mindfulness Based Diet Program on Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Collaborators: Amasya University (Other)
Responsible Party: Principal Investigator, ümüş özbey yücel, Clinical Researcher of the Amasya University Nutrition and Diet Department, Ankara University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AnkaraUniv2
Record Dates: First submitted 2022-04-07; First posted 2022-04-14 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Obesity; Weight Loss
Keywords: Obesity; Weight loss; Mindfulness
MeSH Terms: conditions — Obesity; Weight Loss | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness+Diet intervention (Experimental): Diet and mindfulness intervention
  Interventions: Behavioral: Dietary and mindfulness intervention
- Diet intervention (Experimental): Diet intervention
  Interventions: Behavioral: Dietary and mindfulness intervention

INTERVENTIONS:
Behavioral: Dietary and mindfulness intervention — Dietary intervention: Preparation and follow-up of diet program
  Mindfulness intervention: Implementation of cognitive stress reduction program

SUMMARY:
Meditation interventions, including mindfulness-based approaches, can be effective in reducing psychological stress . Mindfulness meditation, which cultivates awareness of present-moment experience with a nonjudging attitude, is theorized to promote adaptive self-regulation,which is thought to be key to maintaining long-term eating habits and appetite regulation.In the light of this information, in this study, it is aimed to observe the effect of mindfulness approach on body weight and eating behaviours.

DETAILED DESCRIPTION:
The use of minfulness based programs for body weight control and stress management is increasing. One of the main reasons for this situation is that individuals care more about the diet and body weidght as a result of the increase in health concerns and stress. In addition, such cognitive support programs in the diet process provide a more comfortable and stress-free continuation of the diet. Based on the above-mentioned information; in this study, it is aimed to determine the effect of mindfulness based diet intervention on weight loss and eating behaviuors.

Individuals who meet the research criteria will randomize according to their file numbers (with the ramdomizer program) and divide into 2 groups: mindfulness group (15) and control group . Food consumption records, anthropometric measurements and eating behaviours scale of all individuals will record at the beginning and end of the study. In order to prevent interaction between individuals, all diet programs will prepare at different times and individually.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 20-65
* Being obese (BMI≥30 kg/m2)
* Volunteering to participate in research

Exclusion Criteria:

* Being pregnant/lactating
* Having a psychological problem
* Being on a followed diet program

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2022-05-15 (Actual); Primary Completion 2024-06-05 (Actual); Study Completion 2024-07-20 (Actual)

PRIMARY OUTCOMES:
Weight chance | At the end of the 2 months
  BMI (kilogram/ metre2 (kg/m2))

SECONDARY OUTCOMES:
Three factor eating questionnaire (TFEQ) scale score change | At the end of the 2 months
  The score ranges from 0 to 100 points, with an increased score reflecting the eating disorder level

CONTACTS AND LOCATIONS:
Overall Officials: ümüş Ö yücel, Principal Investigator — Ankara University
Locations (1):
- Ümüş Özbey Yücel, Ankara, Select An Option…, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No